CLINICAL TRIAL: NCT02915666
Title: A Phase 1B Clinical Trial of Dabrafenib, Trametinib Plus Digoxin in Patients With Unresectable or Metastatic BRAF V600 Mutant Melanoma
Brief Title: A Clinical Trial of Patients With Melanoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No subjects consented for enrollment on this study.
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 102015-074
Record Dates: First submitted 2016-05-31; First posted 2016-09-27 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Melanoma
Keywords: Melanoma, skin
MeSH Terms: conditions — Melanoma | interventions — digoxin, nicotinic acid, pentifylline drug combination; Digoxin; dabrafenib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Digoxin combination for Melanoma (Experimental): Drugs: Dabrafenib 150mg PO 2x daily, Trametinib 2 mg PO daily, and Digoxin 0.25 mg PO daily for 8-week cycles.
  Interventions: Drug: Digoxin Combination; Drug: Dabrafenib; Drug: Trametinib

INTERVENTIONS:
Drug: Digoxin Combination — Digoxin 0.25 mg PO daily will be given for 8-week cycles
  Other Names: Lanoxin
Drug: Dabrafenib — dabrafenib 150mg PO twice daily for 8-week cycles
  Other Names: Tafinlar
Drug: Trametinib — trametinib 2 mg PO daily for 8-week cycles
  Other Names: Mekinist

SUMMARY:
This study is being done to find out if the combination of dabrafenib, trametinib and digoxin will lessen the side effects that you may experience and to measure your response and duration of response to the combination of drugs.

DETAILED DESCRIPTION:
Melanoma is a cancer of melanocytes--melanin pigment producing cells, and the cancer originates in the skin, uvea, acral tissues and mucosal tissues. Melanoma incidence and mortality are increasing in the U.S. with over 80,000 cases/year and 9,000 deaths/year. Advanced melanoma occurs either after treatment for localized melanoma or de novo and is associated with chemo-resistance and a median survival of 9 months.

The study is a prospective, single-arm, one-site therapeutic trial of the combination of Dabrafenib + Trametinib + Digoxin for advanced V600 mutant melanoma.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic diagnosis of unresectable or metastatic BRAF V600 mutant melanoma.
2. Age > 18 years.
3. Naïve or any number of prior systemic therapeutic regimens for unresectable stage III or stage IV melanoma, except prior BRAF or MEK inhibitor agents. This includes chemotherapy, immunotherapy, biochemotherapy, or investigational treatments. Patients may also have received therapies in the adjuvant setting.
4. Performance status ECOG 0-2.
5. Adequate organ function as defined below:

   A.- total bilirubin 3 x institutional upper limit of normal B.- AST(SGOT)/ALT(SPGT) ≤ 5 X institutional upper limit of normal C.- creatinine 3 mg/dL D.- cardiac ejection fraction > 50% E.- QTcF ≤ 480msec F.-PT/INR/aPTT ≤ 1.5 x institutional upper limit of normal
6. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 4 months following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria: has not undergone a hysterectomy or bilateral oophorectomy; or has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
7. All sites of disease must be evaluated within 4 weeks prior to beginning therapy. Patients must have measurable disease as defined by RECIST v1.1 (see Section 6).
8. Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria

1. Subjects who have had chemotherapy or radiotherapy or any systemic therapy for melanoma within 3 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 3 weeks earlier. No concomitant therapy is allowed including IL2, interferon, ipilimumab, anti-PD-1 or anti-PD-L1 antibody, cytotoxic chemotherapy, immunosuppressive agents, or other investigational therapies.
2. Active infection with hepatitis B or C or HIV.
3. Subjects with active CNS disease are excluded. Patient with brain metastases previously treated with surgery or radiation therapy and with confirmed SD for >2 weeks are allowed.
4. Patients are excluded if they have a history of any other malignancy from which the patient has been disease-free for less than 2 years, with the exception of adequately treated and cured basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix.
5. Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (>class II based on NYHA), unstable angina pectoris, clinically significant and uncontrolled cardiac arrhythmia, uncontrolled thyroid disease, or psychiatric illness/social situations that would limit compliance with study requirements. Acute coronary syndrome within 24 weeks. Note atrial fibrillation controlled >30 days is not an exclusion.
6. History of predisposition to retinal vein occlusion or central serous retinopathy.
7. Prior BRAF or MEK inhibitor therapy.
8. Wolff-Parkinson White syndrome or the presence of an intra-cardiac defibrillator (see Section 7.2.1).
9. Known cardiac metastases.
10. History of interstitial lung disease or unresolved pneumonitis.
11. Immediate or delayed hypersensitivity to digoxin.
12. Patients requiring concomitant medications listed in section 4.3 that are not able to be switched to a reasonable alternative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-07-17 (Actual); Study Completion 2017-07-17 (Actual)

PRIMARY OUTCOMES:
Frequency of DLTs | Every 3 weeks for 36 months
  DLTs will be defined based on the rate of drug-related grade 3-4 toxicities that do not resolve within 3 weeks or any toxicities requiring permanent discontinuation of any of the study drugs

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Frankel, MD, Principal Investigator — UT Southwestern.edu
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No